CLINICAL TRIAL: NCT03032120
Title: Postprandial Response of Fresh-squeezed and Processed Orange Juice on Appetite-related Biomarkers and Antioxidant-status in Lean and Obese Subjects
Brief Title: Postprandial Response of Fresh-squeezed and Processed Orange Juice of Lean and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Thais Cesar, PhD, São Paulo State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SaoPSU17
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fresh orange juice (Experimental): Intervention: The subjects drank 5 mL/kg body weight of fresh-squeezed orange juice (FOJ).
  Interventions: Dietary Supplement: Orange juice
- Processed orange juice (Experimental): Intervention: The subjects drank 5 mL/kg body weight of processed orange juice (POJ).
  Interventions: Dietary Supplement: Orange juice
- Control (Experimental): The subjects drank 5 mL/kg body weight of control drink compounded by water mixed with sugars in a similar concentration of orange juices (5.2% of sucrose, 2.5% of fructose, 2.1% of glucose, 0.75% of citric acid, and malic acid 0.25%, flavored and colored with some drops of orange essence).
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Orange juice — Lean and obese subjects drank one single dose (5 mL/kg body weight) of fresh-squeezed orange juice (FOJ) and processed orange juice (POJ) followed by an ad libitum breakfast. A washout period of seven days among each beverage (FOJ, POJ and control) was applied.
  Arms: Fresh orange juice; Processed orange juice
Dietary Supplement: Control — Lean and obese subjects drank one single dose (5 mL/kg body weight) of an energy and sugars-matched orange-flavored drink (control), followed by an ad libitum breakfast. A washout period of seven days among each beverage (FOJ, POJ and control) was applied.
  Arms: Control

SUMMARY:
This study aimed investigated the acute intake effect of fresh-squeezed orange juice (FOJ), processed orange juice (POJ), and an isoenergetic orange-flavored drink (control) on postprandial response of blood serum biomarkers (glucose, insulin, leptin and adiponectin), anti-oxidatant status, and prospective food intake in lean and obese subjects.

DETAILED DESCRIPTION:
Non-randomized crossover clinical trial, in which eligible participants (n= 36) were allocated in accordance with their body mass index in two groups, lean (n = 18, 9 women/9 men) and obese (n = 18, 9 women/9 men). Subjects of both groups intake of one single dose (5 mL/kg body weight) of isoenergetic beverages in three different phases: (1) fresh-squeezed orange juice (FOJ), (2) commercial processed orange juice (POJ) and (3) an energy and sugars-matched orange-flavored drink (control), with a washout period of seven days among each beverage. Thirty minutes after the intake of each beverage, the participants had a flavonoid-free standard breakfast, which contained coffee (infusion), milk, sugar or sweetener, white bread sandwich with lean ham and light cream cheese, salted and sweet biscuits. Posteriorly, blood samples (10 mL) were collected at 30, 60, 120 and 300 min after each intervention with a catheter installed in a vein of the arm. After blood collection, the volunteers were instructed to record all meals throughout the day, noting the amount eaten of each food. The sample number took into account variations in blood serum glucose with a type I error α = 0.05 and a type II error β = 0.2 (80% power). Primary output were the modification on glucose or insulin concentration induced by different beverages in some point of the curves. The secondary output was the antioxidant activity induced by FOJ and/or POJ. Kolmogorov Smirnov and Levene test, respectively assessed normality and homogeneity of the data. Area under the curve (AUC0-300 min) was calculated by the clearance of the appetite related-biomarkers (glucose, insulin, leptin and adiponectin) during 300 min for each trial phase Other parameters, as maximum concentration (Cmax), and time to reach maximum blood concentration (Tmax) were also estimated. AUC was determined with the trapezoidal method by Microcal Software Inc., Origin® 6.0. One-way analysis of variance (ANOVA) followed by Sidak post hoc was applied to compared the effect of interventions on appetite related-biomarkers, anti-oxidant status and beverage composition. P significance was set up ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women volunteers;
2. Volunteers with BMI between 18.5 to 39.9 kg/m2.

Exclusion criteria:

1. Volunteers with BMI between more than 40 kg/m2;
2. Smokers volunteers;
3. Volunteers who are in treatment with drugs (except contraceptives), vitamins and nutritional supplements;
4. Volunteers who are dieting for weight loss;
5. Volunteers who gained or lost more than 3 kg of weight in the last 3 months;
6. Volunteers who consume more than 20 g of alcohol per day
7. Volunteers who practicing intense physical activity (more than 5 hours per week).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the changes on glucose, insulin, leptin, and adiponectin levels over the time times 0, 30, 60, 120, and 300 min | Up to 6 month after blood collection of glucose, insulin, leptin, and adiponectin.
  Determination of glucose, insulin, leptin, adiponectin in the blood serum.

SECONDARY OUTCOMES:
Assessment of the changes on blood serum antioxidant biomarkers before and after each beverage intervention | Up to 6 month after blood collection of antioxidant biomarkers (TBARS and ABTS).
  Determination of TBARS and ABTS in the blood serum.
Assessing of change on prospective food intake after each beverage intervention | Up to 3 weeks after the application of each 24-h food recall.
  Evaluation of prospective food intake by 24-h food recall.

IPD SHARING:
Plan to Share IPD: No
There was no plan to share individual participant data (IPD) to other researchers.

REFERENCES:
- [Result] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459